CLINICAL TRIAL: NCT05088629
Title: The Relationship of the 3-meter Back Walk Test With Proprioception, Trunk Control and Muscle Strength in Children With Cerebral Palsy
Brief Title: 3-meter Walk Back Test, Proprioception, Trunk Control and Muscle Strength in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sanko University (Other)
Responsible Party: Principal Investigator, zekiye ipek katırcı kırmacı, Asst. Prof., Sanko University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: universitysanko
Record Dates: First submitted 2021-10-11; First posted 2021-10-22 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy; back walk; proprioception; trunk control
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- One group (Other): 3-meter Walk Back Test, Proprioception, Trunk Control and Muscle Strength test
  Interventions: Diagnostic Test: Clinical Tests

INTERVENTIONS:
Diagnostic Test: Clinical Tests — Clinical Tests

SUMMARY:
The gait problems of the child with CP should be examined in detail. At this point, by assigning a different task to the child with the backward walking assessment, body perception, trunk stability provided by anterior-posterior cocontraction, balance, correction and protective reactions are observed. This observation ensures the exact determination of the problem that will guide the treatment.

Back walking is a more difficult activity as it involves neuromuscular control and depends on proprioceptive sense and protective reflexes. In activities of daily living, backward walking is needed to perform tasks such as leaning on a chair and opening the door.

The only test that can be applied to evaluate the ability to walk backwards is the 3 meter back walk test. This test was found to be valid and reliable both in the elderly population and in patients with total knee arthroplasty. In the literature, no study has been found on the factors affecting the three-meter backward walking skills in children with CP. The aim of this study is to examine the relationship between 3 meter back walk test and proprioception, trunk control and muscle strength.

DETAILED DESCRIPTION:
Cerebral palsy is a non-progressive neurodevelopmental disorder that occurs in the immature brain during pregnancy, birth or postpartum. It is the picture of childhood that most frequently causes functional disability. Motor development retardation, balance and posture problems are among the most important problems that cause disability in CP. This picture is often accompanied by cognitive, sensory, perceptual deficiencies, orthopedic disorders and other medical problems. In children with spastic CP, selective movement deficiencies, lack of muscle strength, lack of postural control, lack of proprioception sense, loss of balance and coordination, muscle tone disorders, and motor development delays are seen. Disorders due to muscle tone problems, secondary joint deformations and alignment problems, especially in walking function, are common problems in activities performed against gravity.

Deficiencies in trunk strength and control, lack of strength in antigravity muscles, severity of spasticity, loss of balance and coordination, combined with time-distance problems of walking, cause excessive energy consumption, insufficient for daily living activities and social participation, negatively affecting quality of life, causing muscle and joint problems over time. gait pattern.

The main purpose of the study is to examine the relationship of the 3-meter back walk test with proprioception, trunk control and muscle strength in children with cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

* The age of onset of maturation of walking, in terms of covering the maturation ages and between 6-15 years old,
* Children with CP with a Communication Function Classification System (CFCS) ≤ 3,
* Children with upper extremity muscles ≤ 2 according to the Modified Ashworth Scale (MASH)
* Children in Level-I-II, which are groups with independent walking ability according to Gross Motor Function Classification System,
* Not having any known vision problems in terms of not affecting the postural control responses,
* Not using any pharmacological agent that may affect muscle tone,
* Able to follow verbal commands without mental retardation at a level that interferes with communication,
* Those who have not had any Boutilinum Toxin injection and/or orthopedic surgery in the lower extremity in the last six months,
* Children without epileptic seizures will be included.

Exclusion Criteria:

* Having contractures in any joint of the hip, knee and ankle in the lower extremity,
* Children with hearing and vision problems with any diagnosis will not be included in the study.

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
3 meter back walk test | At baseline
  A distance of three meters will be measured and marked. When the signal is given, they will be asked to walk backwards safely and stop when they reach the marked point.

SECONDARY OUTCOMES:
Proprioception | At baseline
  Evaluation of proprioception with a goniometer
Trunk Control Measurement Scale | At baseline
  It consists of two main parts, static sitting balance and dynamic sitting balance. An increase in the score indicates increased trunk control.
Muscle Strength | At baseline
  Muscle strength will be evaluated with a digital manual muscle dynamometer.
Gillette Functional Walking Assessment Questionnaire | At baseline
  It is an observational assessment scale that evaluates the functional effectiveness of walking.

CONTACTS AND LOCATIONS:
Overall Officials: Nevin ERGUN, Prof., Study Director — Sanko University; Enver KATIRCI, pt, Principal Investigator — Rehabilitation Center; Hatice ADIGÜZEL, asst. prof., Study Director — Kahramanmaras Sutcu Imam University; Zekiye İpek KATIRCI KIRMACI, asst. prof., Study Director — Kahramanmaras Sutcu Imam University
Locations (1):
- Zekiye İpek Katırcı Kırmacı, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Katirci E, Adiguzel H, Katirci Kirmaci ZI, Ergun N. The relationship between the backward walking and proprioception, trunk control, and muscle strength in children with cerebral palsy. Ir J Med Sci. 2023 Oct;192(5):2391-2399. doi: 10.1007/s11845-022-03270-w. Epub 2023 Jan 6. PMID 36604372